CLINICAL TRIAL: NCT05840770
Title: A Phase II Trial of Cemiplimab Alone for Untreated Brain Metastases From PD-L1 ≥ 50% Non-Small Cell Lung Cancer
Brief Title: Cemiplimab for the Treatment of Untreated Brain Metastases From PD-L1 >= 50% Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22346; NCI-2023-02193 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22346 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-05-03 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms | interventions — Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Cemiplimab) (Experimental): Patients receive cemiplimab IV and undergo blood sample collection while on study. Patients undergo MRI, CT scan and PET scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Elastography; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well cemiplimab works in treating patients with PD-L1 >= 50% non-small cell lung cancer (NSCLC) that has spread from where it first started (primary site) to the brain (metastases). Approximately 10% of patients diagnosed with metastatic NSCLC present with brain metastases and another 30% develop brain metastases during the illness. Currently, the management of brain metastases relies on stereotactic radiosurgery (SRS), which has high rates of local control, but in combination with systemic therapy, can cause certain toxicities, including central nervous system (CNS) necrosis or potential cognitive changes or memory deficits. Additionally, in patients with numerous brain metastases, whole brain radiation (WBRT) is recommended, leading to significant neurocognitive deficits. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. However, there is little data on the effectiveness of newer systemic therapies, such as immunotherapy, in penetrating and treating previously untreated brain metastases. Cemiplimab without upfront SRS or WBRT for asymptomatic brain metastases may help delay the need for radiation in patients with untreated brain metastases from PD-L1 >= 50% NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if CNS control rate defined as complete response (CR), partial response (PR), or stable disease (SD), is acceptable with a strategy of cemiplimab alone for patients with advanced NSCLC, PD-L1 >= 50%, no EGFR, ALK or ROS1 aberrations with untreated brain metastases.

SECONDARY OBJECTIVES:

I. To evaluate time until intracranial progression with cemiplimab alone. II. To evaluate time to extracranial progression . III. To evaluate overall survival (OS). IV. To evaluate CNS objective response rate (ORR) defined as CR and PR. V. To evaluate time until administration of radiation therapy (RT), either SRS or WBRT.

VI. To report longitudinal changes in quality of life with cemiplimab alone.

EXPLORATORY OBJECTIVES:

I. To bank blood and tissue specimens for predictive biomarker analyses evaluating CNS disease control and survival outcomes in patients treated with cemiplimab.

OUTLINE: Patients receive cemiplimab intravenously (IV) and undergo blood sample collection while on study. Patients undergo magnetic resonance imaging (MRI), computed tomography (CT) scan and position emission tomography (PET) scan throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Ability to read and understand English for questionnaires
* Histologically confirmed non-small cell lung cancer (NSCLC)
* PD-L1 >= 50%
* Advanced disease
* Measurable disease in the brain >= 1 untreated brain metastasis (measuring 5-15 mm) on brain MRI with contrast within 30 days of enrollment
* Patients must not require corticosteroids for the management of symptoms from their brain metastases in the opinion of the treating investigator
* Patients must be naïve to immune check point inhibitors targeting PD-1 and PD-L1
* Prior treatment with chemotherapy is allowed. Patients who have started chemotherapy for their current disease presentation may have received up to 1 cycle of chemotherapy alone (without cemiplimab) prior to enrollment and the initiation of the protocol-specified regimen of cemiplimab. In patients who have previously received platinum-based chemotherapy for a prior disease presentation, for eligibility there must be at least 21 days since the last exposure to platinum-based chemotherapy
* Prior exposure to immune checkpoint inhibitors targeting PD-1 and/or PD-L1 is allowed if patients have been off of therapy for at least 1 year Life expectancy >= 3 months in the opinion of the treating investigators
* Up to 10 asymptomatic (defined as no neurologic symptoms at presentation and not requiring steroids) brain lesions allowed up to 15 mm in size. Patients with lesions > 15 mm or with a lesion at or near a critical structure (i.e. brainstem, optic structures) may still be eligible if that lesion(s) is treated and others are available that fit the above criteria
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 30 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 1.5 x ULN (performed within 30 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 3 x ULN (performed within 30 days prior to day 1 of protocol therapy)
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 30 days prior to day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 30 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* No EGFR, ALK or ROS1 aberrations
* Brainstem lesion or threatening lesion adjacent to critical structures (i.e. optic nerves/chiasm) - patients can still be enrolled if these are treated and additional lesion(s) based on inclusion criteria above are met
* Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months; patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study; subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study; subjects with hypothyroidism stable on hormone replacement are not excluded from this study
* Has had a prior monoclonal antibody within 4 weeks or 5 half-lives, whichever is shorter, prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy or targeted small molecule therapy within 3 weeks prior to administration of the study drug or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent;

  * Note: Subjects with permanent =< grade 2 toxicities (e.g. neuropathy) or toxicities corrected through routine medical management (e.g. thyroid replacement for hypothyroidism), are an exception to this criterion and may qualify for the study;
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy; *Note: Subjects with =< grade 2 amylase or lipase elevations abnormalities that have no corresponding clinical manifestations (e.g. manifestation of pancreatitis), are an exception to this criterion and may qualify for the study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, indolent lymphomas, or in situ cervical cancer that has undergone potentially curative therapy or any additional tumor that has been deemed to be effectively treated with definitive local control (with or without continued adjuvant hormonal therapy) for at least 2 years prior to enrollment
* Prior whole brain radiation
* Has known carcinomatous meningitis (also known as leptomeningeal disease)
* Is taking > 4mg/day of dexamethasone or its equivalent at the start of immunotherapy or has required > 4mg/day of dexamethasone or its equivalent for 3 consecutive days within 1 week of starting treatment
* > 10 brain metastases
* Patients whose tumor exhibit activating EGFR mutation, ALK or ROS translocation and have a standard of care molecular targeted therapy available for these mutations, will be excluded from this study; adenocarcinoma patients may be consented prior to the EGFR and ALK status being known, but EGFR and ALK status must be determined prior to initiating therapy
* Previous CNS surgery within 2 weeks of treatment, with the exception of biopsy
* Unable or unwilling to undergo an intracranial MRI
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS) control rate | At 4 weeks
  Includes complete response (CR), partial response (PR), and stable disease (SD) using Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Time until any CNS progression | Up to 12 months from time of enrollment
  Measured by RANO-BM criteria .
Extracranial progression free survival | From enrollment to progression or death due to any cause, assessed up to 2 years
  Defined as first occurrence of disease progression by Positron Emission Response Criteria in Solid Tumors version (v) 1.0 or Response Evaluation Criteria in Solid Tumors v1.1.
Time until administration of whole brain radiation therapy or stereotactic radiosurgery | Up to 5 years
Incidence of adverse events | Up to 2 years
  Rate of all grades and grade >= 3 toxicities at least possibly related to study therapy as measured by Common Terminology Criteria for Adverse Events v 5.0.
Overall survival | From the date of study enrollment to the date of death from any cause, assessed up to 5 years
Time until brain metastases-specific mortality | Up to 24 months from enrollment
  Defined as intracranial progression as a component of cause of death per RANO-BM criteria.
Cumulative rate of best responses | Up to 5 years
  Individually for CR, PR, SD as defined by the RANO-BM criteria.
Longitudinal changes in patient-reported quality of life - Measurement I | Baseline to day 42
  Measured by using the MD Anderson Symptom Inventory-Brain Tumor, Patient-Reported Outcomes Measurement Information System Cognitive Function Short Form (4a), and linear analogue self-assessment single-item numerical scale.MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT): scale of 0 (not present) - 10 (as bad as you can imagine). 28 questionnaire with minimum score of 0 (best score) and maximum score of 280 (worse score).
Longitudinal changes in patient-reported quality of life - Measurement II | Baseline to day 42
  Measured by using Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function Short Form. Scale of 5 (never) - 1 (very often/several times a day). 6 questions with a minimum score of 6 (worse score) and maximum score of 30 (best score).
Longitudinal changes in patient-reported quality of life - Measurement III | Baseline to day 42
  Measured by using Linear Analogue Self-Assessment (LASA) Single-Item Numerical Scale. Scale of 0 (as bad as it can be) - 10 (as good as it can be). 5 questions with a minimum score of 0 (worse score) and maximum score of 50 (best score).

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center